CLINICAL TRIAL: NCT07376538
Title: A Prospective Phase II Clinical Study of Response-Based Local Therapy After Systemic Therapy in Regionally Advanced Breast Cancer
Brief Title: Response-Based Local Therapy for Regionally Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang,MD, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5176
Record Dates: First submitted 2026-01-20; First posted 2026-01-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Regionally Advanced Breast Cancer; Hypofractionated Radiotherapy; Systemic Consolidation Therapy; Breast Surgery; Regional Lymph Node Dissection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Response-Adapted comprehensive treatment strategy (Experimental)
  Interventions: Radiation: Response-adapted comprehensive treatment strategy

INTERVENTIONS:
Radiation: Response-adapted comprehensive treatment strategy — Participants will receive a response-adapted comprehensive treatment strategy following neoadjuvant systemic therapy (NST). The strategy includes:
  Surgery: Patients with residual ISLN/IMLN ≥ 0.5 cm after NST are assigned (1:1) to receive either regional lymph node dissection or no dissection, in addition to standard breast and axillary surgery.
  Radiotherapy: Patients receive individualized, dose-adaptive hypofractionated or conventional fractionation radiotherapy guided by the response of the breast and regional nodes to NST.
  Systemic Therapy: Intensified consolidation systemic therapy is administered based on NST efficacy.

SUMMARY:
The goal of this interventional clinical trial is to evaluate if an individualized treatment strategy (involving radiation boost, surgery, and systemic consolidation) can improve progression-free survival in patients with breast cancer presenting with positive ipsilateral supraclavicular (ISLN) and/or internal mammary lymph nodes (IMLN).

The main questions it aims to answer are:

Is individualized hypofractionated radiotherapy with a local boost safe and effective when adjusted by the response to neoadjuvant treatment?

Does local surgery provide benefit for patients who have high residual tumor burden in these lymph nodes after neoadjuvant treatment?

How effective is intensified systemic therapy when tailored to the patient's molecular subtype?

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 to 75 years.

ECOG performance status ≤ 2.

Histologically confirmed invasive breast cancer.

Newly diagnosed breast cancer with pathologically confirmed positive ipsilateral supraclavicular lymph nodes (ISLN) and/or internal mammary lymph nodes (IMLN); for patients in whom IMLN biopsy is not feasible, clinically positive IMLN based on investigator assessment and imaging findings is acceptable.

Planned to receive neoadjuvant systemic therapy followed by breast-conserving surgery or mastectomy and axillary lymph node dissection, with or without supraclavicular and/or internal mammary lymph node dissection.

Adequate baseline organ function, defined as: absolute neutrophil count ≥ 1.5 × 10⁹/L; platelet count ≥ 100 × 10⁹/L; hemoglobin ≥ 9 g/dL (90 g/L); serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min; total bilirubin ≤ 1.5 × ULN; AST and/or ALT ≤ 2.5 × ULN; INR ≤ 1.5 and PT/APTT ≤ 1.5 × ULN.

Able and willing to comply with study procedures and scheduled follow-up.

Written informed consent obtained prior to any study-related procedures.

Exclusion Criteria:

Evidence of distant metastatic disease.

Presence of severe or uncontrolled concomitant diseases, including severe cardiac dysfunction; myocardial infarction, uncontrolled arrhythmia, or unstable angina within 3 months prior to enrollment; clinically significant pericardial disease; or severe pulmonary disease.

Prior radiotherapy to the chest wall or supraclavicular region.

Pregnancy, lactation, or any condition considered by the investigator to contraindicate radiotherapy.

History of or concurrent second primary malignancy, except for non-melanoma skin cancer, papillary or follicular thyroid carcinoma, carcinoma in situ of the cervix, contralateral non-invasive breast cancer, or other malignancies treated with curative intent with no evidence of disease for more than 3 years.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 157 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
Cumulative Incidence of Locoregional Recurrence | Up to 5 years
Cumulative Incidence of Distant Metastasis | Up to 5 years
Incidence of Treatment-Related Toxicities | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No